CLINICAL TRIAL: NCT05745987
Title: SMART (Smallpox Vaccine for Mpox Post-Exposure Prophylaxis: A Cluster Randomized Controlled Trial)
Brief Title: Smallpox Vaccine for Mpox Post-Exposure Prophylaxis: A Cluster RCT
Acronym: SMART
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMART RCT
Record Dates: First submitted 2023-02-10; First posted 2023-02-27 (Actual); Last update posted 2025-07-06 (Actual); Status verified 2025-07

CONDITIONS: Monkeypox
Keywords: mpox
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Intervention Model Description: Each group will be randomly selected to receive the smallpox vaccine or the typhoid vaccine
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not know which vaccine they receive until after the study is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smallpox vaccine (Experimental): Participants will receive the Bavarian Nordic smallpox vaccine 0.5 ml single-dose
  Interventions: Drug: Bavarian Nordic smallpox vaccine
- Typhoid vaccine (Active Comparator): Participants will receive the Typhim Vi® typhoid vaccine 0.5 ml single-dose
  Interventions: Drug: Typhoid VI Polysaccharide Vaccine Injectable Solution

INTERVENTIONS:
Drug: Bavarian Nordic smallpox vaccine — A single dose of the Bavarian Nordic smallpox vaccine will be given at baseline.
  Other Names: Imvamune
  Arms: Smallpox vaccine
Drug: Typhoid VI Polysaccharide Vaccine Injectable Solution — A single dose of the typhoid vaccine will be given at baseline.
  Arms: Typhoid vaccine

SUMMARY:
A cluster randomized controlled trial to determine if smallpox vaccine reduces secondary cases and symptom severity in persons exposed to mpox.

DETAILED DESCRIPTION:
A pragmatic, adaptive, multi-site, cluster randomized trial where households with one or more persons confirmed to have mpox will be randomized to smallpox vaccine or control. The co-primary outcomes are RT-PCR confirmed mpox and symptom severity.

ELIGIBILITY:
Inclusion Criteria:

1. Household member of person with laboratory confirmed mpox
2. Age ≥ 2 years
3. Within 14 days of onset of illness in mpox index case

Exclusion Criteria:

1. Pregnancy
2. Breastfeeding
3. Past serious allergic reaction to study vaccine components
4. Previous smallpox vaccination
5. Current or planned use of another investigational drug at any point during study participation

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
PCR-confirmed Mpox | 8 weeks
  To evaluate if smallpox vaccine vs control prevents RT-PCR confirmed mpox
Symptom severity | 8 weeks
  To evaluate if smallpox vaccine vs control affects symptom severity

SECONDARY OUTCOMES:
Resolution of skin lesions | 8 weeks
  To assess the time to resolution (i.e. a new skin layer has formed) of any skin lesion
Number of skin lesions | 8 weeks
  To assess the number of skin lesions for any participants who develop mpox
Self-reported Quality of Life | 8 weeks
  To assess the QOL of participants using the World Health Organization Quality of Life Scale
Mpox complications | 8 weeks
  To assess longitudinal complications for any participants who develop mpox
Mpox Pain | 8 weeks
  To assess pain using an adapted Zoster Brief Pain Inventory
Hospitalization | 8 weeks
  To determine all cause hospitalization over the study period
Mortality | 8 weeks
  To determine all cause mortality over the study period

OTHER OUTCOMES:
Safety (SAEs, AESI) | 6 months
  Solicited SAE and AESIs will be followed at 4 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, Principal Investigator — McMaster University
Locations (10):
- Catholic University of Bukavu, Kinshasa, Bukavu, Democratic Republic of the Congo
- Nigeria (8):
  - Federal Medical Center, Abuja
  - University of Abuja Teaching Hospital, Abuja
  - University of Ibadan, Ibadan
  - Irrua Specialist Teaching Hospital, Irrua
  - Aminu Kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos
  - Niger Delta Teaching Hospital, Okolobiri
  - University of Port Harcourt Teaching Hospital, Port Harcourt
- Makerere University Lung Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No